CLINICAL TRIAL: NCT06799130
Title: Effect Of Instrument-Assisted Soft Tissue Mobilization Versus Muscle Energy Technique Over Sternocleidomastoid In Patients With Chronic Non-Specific Neck Pain
Brief Title: Instrument-Assisted Soft Tissue Mobilization Versus Muscle Energy Technique on Chronic Non-specific Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, alaa mohamed hassan saleh, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005583
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: CHRONIC NON-SPECIFIC NECK PAIN
Keywords: instrument-assisted soft tissue mobilization; muscle energy technique

STUDY DESIGN:
Intervention Model Description: instrument assisted soft tissue mobilization and muscle energy technique
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- instrument-assisted soft tissue mobilization (Experimental): the patients will receive instrument-assisted soft tissue mobilization twice a week for four weeks over sternocleidomastoid muscle bilaterally utilizing an M2T blade. The subject lay comfortably in supine position on a treatment table. After using alcohol swabs to clean the patient's skin and the blade, a lubricant (Vaseline) will be applied, and a sweeping technique will be utilized to administer a thorough yet comfortable soft tissue mobilization on the sternocleidomastoid from origin to insertion for roughly 3 minutes.
  conventional therapy the patients will receive hot back for 15 minutes, neck range of motion (ROM), chin tuck, stretches and strengthen exercise.
  Interventions: Other: instrument-assisted soft tissue mobilization; Other: Muscle energy technique
- Muscle energy technique (Experimental): the patients will receive post-isometric muscle relaxation(PIR) treatment for the sternocleidomastoid muscle, it will be applied from supine lying position with the head free from the plinth and held by the therapist's hand, the therapist placed one hand opposite the side of involvement muscle , The other hand is placed on the involved side of muscle . The patient pushed upward against the therapist's thumb on the forehead and looked up, then the patient will be asked to stop pushing and look down. After relaxation therapist will stretch the muscle for 30 seconds. This will be repeated 3 times bilaterally for 3 sessions per week for four weeks.
  conventional therapy the patients will receive hot back for 15 minutes, neck range of motion, chin tuck, stretches and strengthen exercise.
  Interventions: Other: instrument-assisted soft tissue mobilization; Other: Muscle energy technique
- conventional therapy (Active Comparator): the patients will receive conventional therapy three times a week for four weeks conventional therapy the patients will receive hot back for 15 minutes, neck range of motion (ROM), chin tuck, stretches and strengthen exercise.
  Interventions: Other: instrument-assisted soft tissue mobilization; Other: Muscle energy technique

INTERVENTIONS:
Other: instrument-assisted soft tissue mobilization — instrument-assisted soft tissue mobilization
  Other Names: IASTM
Other: Muscle energy technique — Muscle energy technique

SUMMARY:
the aim of this study is to investigate if there is any difference between INSTRUMENT-ASSISTED SOFT TISSUE MOBILIZATION and Muscle Energy Technique over sternocleidomastoid on Neck pain, Range of motion and Functional disability in patients with Chronic Non-specific Neck Pain

DETAILED DESCRIPTION:
Non-specific neck pain (NSNP) is the most common and the 4th leading cause of musculoskeletal disorder worldwide. It is estimated that about 70% of the population experiences neck pain throughout life, with an annual incidence of 15% to 50%0. It is seen more commonly in middle-aged females. It has been well established that NSNP is not only the risk factor for developing severe spinal pathologies and functional disability but that it is also associated with decreasing the quality of life and productivity of workers. Pain, which leads to functional limitations especially in the cervical region, is associated with a decrease in the activation of the deep cervical flexors such as the longus colli and longus capitis muscles, and an increase in the activation of the superficial cervical flexors, such as SCM and anterior scalene muscles.It is reported that in individuals with CNP, there is an increase in the activation of SCM and anterior scalene muscles, especially during isometric cervical flexion and dynamic upper limb movements. In their study, Falla et al. concluded that individuals with unilateral CNP had muscle fatigue in their ipsilateral SCM and anterior scalene muscles. Wang et al. reported postural imbalance in individuals with CNP due to an increased activation and tightening of the suboccipital, SCM, upper trapezius, pectoralis, and rotator cuff muscles. A study by Mostafa et al., (2021) stated that IASTM has a favorable effect than conventional treatment in reduction mechanical neck pain, improvement cervical range of motion &activity of daily living.

A Systematic Review by Sbardella et al., (2021) stated that all the studies analyzed show an effective improvement in the outcomes of pain, disability and joint function, which leads us to say that Muscle Energy Technique (MET) is certainly an effective and safe technique in the treatment of cervical pain.

this trail has three groups; one will receive IASTM+ conventional, the second will receive Muscle energy technique+ conventional and the third one will receive conventional treatment for four weeks

ELIGIBILITY:
Inclusion Criteria:

1. The subjects are of both genders, aged between 18-35 years old .
2. Subjects with Neck pain continued for at least the last 12 weeks .
3. body mass index (18.5-24.9).

Exclusion Criteria:

1. Any specific neck pathology as radiculopathy, rheumatoid arthritis, and systemic diseases
2. Sensory problems at the mid or upper back .
3. A tendency to hemorrhage or anticoagulation treatment. And nonsteroidal pain medication .
4. Signs of severe pathology such as malignancy, fractures of the cervical spine, cervical radiculopathy or myelopathy, or vascular syndromes such as vertebrobasilar insufficiency .
5. surgery of the cervical spine, whiplash trauma (in the past or recent, as cause of the complaint).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-29 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to four weeks
  the scale that will be used is VAS ; each subject will be instructed to put point on line from no pain to tolerable pain

SECONDARY OUTCOMES:
neck range of motion | up to four weeks
  will be measured by cervical range of motion device (CROM)
neck disability | up to four weeks
  will be measured by Arabic version of neck disability index

CONTACTS AND LOCATIONS:
Overall Officials: alaa saleh, Principal Investigator — Cairo University
Locations (1):
- Alaa Mohamed Hassan Saleh, Cairo, Egypt